CLINICAL TRIAL: NCT02247102
Title: Placebo-controlled Randomized Trial to Investigate the Breath Hydrogen Exhalation After a Test Meal Containing Isomaltulose (Palatinose™) or Sucrose in Infants Aged 6-12 Months
Brief Title: Investigate the Breath Hydrogen Exhalation After a Test Meal Containing Isomaltulose or Sucrose in Infants
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Beneo GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: TASMC-14-NV-132-CTIL
Record Dates: First submitted 2014-09-19; First posted 2014-09-23 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Malabsorption
MeSH Terms: conditions — Malabsorption Syndromes | interventions — isomaltulose; Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isomaltulose (Experimental): Dosage of 1 g/ kg body weight (rounded up to the nearest 0.5 kg)
  Interventions: Dietary Supplement: Isomaltulose; Dietary Supplement: Sucrose
- Sucrose (Active Comparator): Dosage of 1 g/ kg body weight (rounded up to the nearest 0.5 kg)
  Interventions: Dietary Supplement: Isomaltulose; Dietary Supplement: Sucrose

INTERVENTIONS:
Dietary Supplement: Isomaltulose — Each subject receives isomaltulose on Study Day 1. After having completed the wash-out period, each subject receives sucrose on Study Day 2.
  Dosage of 1 g/ kg body weight (rounded up to the nearest 0.5 kg).
  Other Names: Palatinose™
Dietary Supplement: Sucrose — Each subject receives sucrose on Study Day 1. After having completed the wash-out period, each subject receives isomaltulose on Study Day 2.
  Dosage of 1 g/ kg body weight (rounded up to the nearest 0.5 kg).

SUMMARY:
The study shall investigate whether isomaltulose

* is digested and absorbed to a comparable degree like other carbohydrates (CHO) used as ingredients for this age group (e.g. sucrose), by measuring the H2 exhalation in the postprandial period
* does not mediate abdominal discomfort or diarrhoea and is therefore as well tolerated as other CHO (e.g. sucrose), by/in healthy infants aged 6 to 12 months.

It is hypothesized that isomaltulose, provided with a standard follow-on formula,

1. will not significantly increase the mean basal breath H2-excretion rate (determined as the incremental area under the curve (iAUC) of H2-exhalation) over a 3 h postprandial period compared to a sucrose containing standard follow-on formula.
2. will not lead to a significantly different gastrointestinal tolerance in the conse-quent 24 h after formula consumption compared to a sucrose containing standard follow-on formula in infants aged 6 to 12 months.

DETAILED DESCRIPTION:
The intervention will be scheduled on Study Day 1 and Study Day 2. The caretakers will be asked to feed their infant with their usual standard formula in the morning of Study Day 1 and Study Day 2 at home (at their regular feeding time). At the study center, the infant will consume his usual follow-up formula in the usual amount to wich the study product (palatinose or sucrose 1 gram/kg body weight) will be added to the nearest 0.5 kg weight. The introduction will be in the second meal of the day and the time between the first feeding and the interventionwill be of 4h. Before and after the single consumption of the study formula (baseline vs. test condition), the H2 exhalation of the infant will be measured and monitored every 30 min for an additional period of 3 h. In between Study Days 1 and 2, a wash-out period of at least 2 days will be implemented to reduce the potential occurrence of carry-over effects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject was healthy-born at term (37th-42th gestational week) and is healthy at the time of pre-examination
2. Subject is aged 6-12 months at the time of pre-examination
3. Subject ranges between 5th and 95th percentile for age (EURO Growth Guide-lines)
4. Subject has been formula-fed (and complementary food, such as fruit or car-rots, have already been introduced) and not exclusively breast-fed for at least 4 weeks prior onset of the trial
5. Parents/caretakers understand the English or Hebrew language and are able and willing to follow the study instructions and fill out questionnaires
6. Subject is suitable for participation in the study according to the PI/study per-sonnel
7. Parents/caretakers have voluntarily agreed to participate and successfully completed the informed consent form (ICF)

Exclusion Criteria:

1. Subject is a pre-term (<37th gestational week)
2. Subject or mother is suffering from an acute or chronic disease followed by medication therapy at the time of pre-examination
3. Subject is suffering from (congenital) gastrointestinal disease or malformation (followed by medication)
4. Subject is suffering/ suffered from infection (which lead to diarrhoea or vomit-ing) in previous 14 days
5. Subject has been administered antibiotics and/or laxatives in the previous 14 days prior to the start of the intervention
6. Subject has a (hereditary) fructose/lactose intolerance and/or (food) allergy
7. Subject is suffering from carbohydrate malabsorption
8. Drug or alcohol abuse by mother of subject
9. Subject is a hydrogen non producer.
10. Subject is currently involved or will be involved in another clinical or food study
11. Subject is not suitable for participation in the study according to the PI/study personnel
12. It is impossible for the subject to travel to the study center on Study Days 1 and 2

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-02 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
hydrogen breath | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nachum Vaisman, MD, Principal Investigator — The Tel Aviv Sourasky Medical Center
Locations (1):
- The Tel Aviv Sourasky Medical Center, Tel Aviv, Israel